CLINICAL TRIAL: NCT00065299
Title: Effects of Maternal Phenylketonuria (PKU) on Pregnancy Outcome
Brief Title: Low Phenylalanine Diet for Mothers With Phenylketonuria (PKU)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-PKU; 1N01HD23148; 1N01HD23155; 1N01HD23156
Record Dates: First submitted 2003-07-21; First posted 2003-07-22 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-05

CONDITIONS: Phenylketonuria
Keywords: Hyperphenylalaninemia; PKU; Maternal PKU; Pregnancy outcome; Phenylalanine restricted diet; Tyrosine supplementation; Maternal hyperphenylalanemia during pregnancy
MeSH Terms: conditions — Phenylketonurias; Phenylketonuria, Maternal

INTERVENTIONS:
Behavioral: Restricted phenylalanine diet

SUMMARY:
Phenylketonuria (PKU) is a rare genetic condition. If not treated, PKU can cause severe mental retardation. Women with PKU are advised to eat a special diet when pregnant to prevent mental retardation in their children. This study will evaluate the effects of that diet on the children of mothers with PKU.

DETAILED DESCRIPTION:
PKU is an autosomal recessive trait caused by the absence of phenylalanine hydroxylase. Phenylalanine hydroxylase is an enzyme involved in the metabolism of phenylalanine (Phe). When phenylalanine hydroxylase is absent or defective, Phe levels rise and toxic Phe metabolites accumulate, causing central nervous system injury. PKU is a treatable disease. Affected individuals must adhere to a diet low in Phe during childhood. Women with PKU should also adhere to a low Phe diet before and during pregnancy to avoid fetal damage. The offspring of women with untreated maternal hyperphenylalaninemia (HPA) usually exhibit mental retardation, microcephaly, growth retardation, and other congenital anomalies. This study will examine the effect of a restricted Phe diet on reproductive outcome in women with maternal HPA.

Participants in this study will be women with HPA whose blood Phe values are persistently greater than 4 mg/dl. Those women with blood Phe values consistently greater than 8 mg/dl will be placed on a Phe restricted diet to maintain plasma Phe concentrations between 2 and 8 mg/dl. This level of control is practical and achievable. Due to a gradient of increasing Phe level from mother to fetus, levels in the latter would vary from 3.5 to 12 mg/dl; these levels are usually associated with normal outcomes. Women will be monitored throughout their pregnancy on obstetric, biochemical, and nutritional parameters. Women on the Phe restricted diet will be given enough Phe-limited protein, calories, vitamins, and minerals to maintain adequate nutritional status. Folate supplementation will be provided. If indicated clinically, tyrosine (Tyr) and supplemental trace metals will be prescribed.

A matching control sample of women and their offspring will be developed in collaboration with associated coordinating and collaborating centers. The offspring of both groups of mothers will be followed as long as the project permits. Those offspring born to mothers admitted to the project during the first 2 to 3 years of the study will be assessed on their intellectual ability and physical health, as well as academic achievement in school. Those admitted during the last 3 to 4 years of the study will be assessed on their intellectual ability and physical health, recognizing that limited data will be available for these offspring.

ELIGIBILITY:
Inclusion Criteria

* Live in community setting
* Become pregnant or give birth during the term of the investigation
* Identified early in pregnancy
* Dietary therapy instituted prior to conception whenever possible
* Diagnosis of PKU based on results of Phe challenge, or clear diagnostic evidence in medical record
* Blood Phe > 4 mg/dl
* Intellectually able to understand and comply with the requirements of the Phe restricted diet, understand an informed consent, and adequately communicate with clinic personnel
* IQ > 70

Inclusion Criteria for Controls

* Heterozygous sisters to HPA women
* Matched control from maternity facility; pregnancy and offspring from a non-PKU female and a PKU male

Exclusion Criteria

* Women with evidence of pterin defect

Min Age: 0 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 572
Dates: Start 1984-05; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Richard Koch, M.D., Principal Investigator — University of Southern California; Reuben Matalon, M.D., Principal Investigator — University of Illinois at Chicago; Bobbye M. Rouse, M.D., Principal Investigator — University of Texas at Galveston
Locations (3):
- United States (3):
  - University of Southern California School of Medicine, Los Angeles, California
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Texas Medical Branch at Galveston, Galveston, Texas

REFERENCES:
- [Background] Levy HL, Guldberg P, Guttler F, Hanley WB, Matalon R, Rouse BM, Trefz F, Azen C, Allred EN, de la Cruz F, Koch R. Congenital heart disease in maternal phenylketonuria: report from the Maternal PKU Collaborative Study. Pediatr Res. 2001 May;49(5):636-42. doi: 10.1203/00006450-200105000-00005. PMID 11328945
- [Background] Koch R, Levy HL, Matalon R, Rouse B, Hanley WB, Trefz F, Azen C, Friedman EG, de la Cruz F, Guttler F, et al. The international collaborative study of maternal phenylketonuria: status report 1994. Acta Paediatr Suppl. 1994 Dec;407:111-9. doi: 10.1111/j.1651-2227.1994.tb13468.x. PMID 7766945
- [Background] Matalon R, Michals K, Azen C, Friedman E, Koch R, Rouse B, Hanley WB, de la Cruz F. Maternal PKU Collaborative Study: pregnancy outcome and postnatal head growth. J Inherit Metab Dis. 1994;17(3):353-5. doi: 10.1007/BF00711828. No abstract available. PMID 7807951
- [Background] Koch R, Levy HL, Matalon R, Rouse B, Hanley W, Azen C. The North American Collaborative Study of Maternal Phenylketonuria. Status report 1993. Am J Dis Child. 1993 Nov;147(11):1224-30. doi: 10.1001/archpedi.1993.02160350098015. PMID 8237918
- [Background] Koch R, Hanley W, Levy H, Matalon R, Rouse B, Dela Cruz F, Azen C, Gross Friedman E. A preliminary report of the collaborative study of maternal phenylketonuria in the United States and Canada. J Inherit Metab Dis. 1990;13(4):641-50. doi: 10.1007/BF01799519. PMID 2122127